CLINICAL TRIAL: NCT01160900
Title: Phase III Study, Multivessel Percutaneous Treatment During Myocardial Infarction
Brief Title: FIT (Fast Infarction Treatment): Complete Revascularization During Primary Percutaneous Coronary Intervention (PCI) Can be Achieved Safely With an Improved Clinical Outcome During the Indexed Hospitalization.
Acronym: FIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Interventional Cardiology, A O San Camillo Forlanini Rome, Marco Stefano Nazzaro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sperimental Registry n°844
Record Dates: First submitted 2010-07-06; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Myocardial Infarction; Ischemia; Heart Failure; Necrosis; Stents
Keywords: cardiovascular diseases; heart disease; hemorrhage; coronary angioplasty; drug eluting stents
MeSH Terms: conditions — Myocardial Infarction; Ischemia; Heart Failure; Necrosis; Cardiovascular Diseases; Heart Diseases; Hemorrhage | interventions — Drug-Eluting Stents; Prasugrel Hydrochloride; bivalirudin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- multivessel revascularization (Experimental): Complete Revascularization : the Infarcted related artery was opened followed by dilatation of other significantly narrowed arteries during the same procedure
  Interventions: Procedure: Coronary angioplasty all lesions

INTERVENTIONS:
Procedure: Coronary angioplasty all lesions — treatment by coronary angioplasty and drug eluting stent of all lesions, adjunctive use of prasugrel and bivalirudin
  Other Names: drug eluting stent, prasugrel, bivalirudin

SUMMARY:
Few reports described outcomes of complete compared with infarct related artery (IRA) only revascularization in patients with ST elevation myocardial infarction (STEMI) and multivessel coronary disease (CAD).

The purpose of this study is to determine outcome (death, myocardial infarction, target vessel failure) of 180 consecutive patients with STEMI and multivessel CAD undergoing primary angioplasty.

Before the first angioplasty patients are randomized to 2 different strategies: 1) culprit vessel angioplasty only, 2) staged revascularization.

ELIGIBILITY:
Inclusion Criteria:

* myocardial acute infarction
* prolonged chest pain (>20 minute) started less <12 hours before arrive in hospital
* ST segment elevation of >1mm in >2 contiguous leads
* new left bundle branch block
* diameter of the coronary suitable of angioplasty >2mm
* the patients agrees to the study protocol and provides a written consensus
* two or more coronary suitable for angioplasty

Exclusion Criteria:

* refused written consensus
* hypersensitivity or contraindication to any of the following medications: heparin bivalirudin aspirin prasugrel stainless steel
* history of bleeding
* cardiogenic shock (PA < 90mmHg)
* chronic total occlusion in the second lesion
* TIMI Flow < II in the culprit lesion
* recent pregnancy
* history of intra-cerebral major hemorrhagic stroke
* an elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first six months post enrollment life expectancy <1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
death at 30 days | 1 month
stent thrombosis | 1 year
target vessel failure | 1 year
re-acute myocardial infarction | 1 month

SECONDARY OUTCOMES:
bleeding | 1 month
timi frame count | 1 day
vascular site access complications | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera San Camillo Forlanini, Roma, Italy, Italy